CLINICAL TRIAL: NCT04465604
Title: HYPERTONIC SALINE COATED FACE MASK FOR REDUCING RESPIRATORY SYMPTOM SEVERITY IN PATIENTS WITH COVID-19
Brief Title: Hypertonic Saline for COVID-19 Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC # 2201072; H-01-R-007 (Other: NCBE Registration (KSA))
Record Dates: First submitted 2020-07-02; First posted 2020-07-10 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: The sample size was based on the following assumptions: Poor response rate to HTS is set at 10% or less; Good response to HTS is set at 30% or more ;One-sided Alph error probability is set to < 0.05 (i.e. p < 0.05) and Power to detect rate difference between good response and poor response to HTS is at least 80%. Using the Fleming single-arm group-sequential design (Fleming 1982) Based on these assumptions; a sample size of N=25 patients is expected to achieve a power of 84% of detecting enough activity by HTS (p<0.05 one-sided) of improving respiratory parameters of COVID19 patients. This will be achieved if the true remission rate difference between a poor and good HTS is 20%. Considering the dropout rate of 25%, a minimum of 50 patients will be enrolled. This will ensure more than 90% power to detect at least 20% positive effect of HTS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Wearing surgical face mask sprayed with hypertonic saline — The inner surface of a standard surgical face mask will sprayed by 10 to 15 ml of HTS (6% w/v Saline solution prepared by adding 6 gram NaCl to 100 ml of water if not commercially available) and allowed to air dry. The participant will wear the face mask for 20-30 minutes every 6 hours until discharge, intubation for mechanical ventilation or death. A new HTS sprayed mask will be worn by the participant every 24 hours. The data items will be collected on daily basis

SUMMARY:
Rationale:

Coronavirus disease 2019 (COVID-19) is spreading rapidly in the world with no proven effective therapy to date. Some patients with COVID-19 develop sever respiratory disease requiring ICU care. There is in vitro evidence that hypertonic saline (HTS) may be beneficial in reducing the inflammatory component in similar viral illnesses.

Objective:

To assess whether wearing a face mask sprayed with HTS (in addition to other COVID-19 treatments) leads to decreasing the severity of the respiratory symptoms resulting from COVID-19.

Study design:

Multi-centre trial

Study population:

Any patient older than 18 years of age with confirmed COVID-19 diagnosis who has any of the following respiratory symptoms or signs:

* cough,
* shortness of breath,
* tachypnea (respiratory rate of 20 breaths / minute or more),
* hypoxemia (O2 saturation 90% or less on room air)

Intervention:

Participants will be asked to wear a face mask for 20-30 minutes every 6 hours for the duration of their respiratory symptoms and/or signs. This inside surface of the face mask will be sprayed with 10-15 ml of HTS and allowed to air dry before the participant is permitted to wear it. A new face mask will be given to the patient every 24 hours. All participants will continue to receive their other COVID-19 treatments as per local hospital guidelines.

Main study parameter:

Improvement of the respiratory symptoms and signs on repeated measurement.

Nature and extent of the burden and risks associated with participation, benefit:

The burden of COVID-19 is very severe world wide. The trial duration is 3 months, with potential extension if deemed needed by interim analysis at the end of 3 months. There are no additional risks for participation in this study as only face masks will be used with no additional medications being given to the participants. In the future, the results of this study could lead to improved care for COVID-19 patients.

DETAILED DESCRIPTION:
Since its emergence as severe outbreak in China in December 2019, coronavirus disease 2019 (COVID-19) has spread so rapidly in the world that more than 780,000 cases have so far been reported worldwide and since then the WHO has declared it as a pandemic. The rapid spread of the disease is imposing major threats on healthcare systems in many countries in the world The major threat to these healthcare systems so far has been the large number of patients who will need respiratory support (ventilators) because of the severe lung injury associated with COVID-19.This disease shares similar pathogenetic, epidemiological and clinical features to the two previously reported coronavirus epidemics (severe acute respiratory syndrome [SARS] and Middle East respiratory syndrome [MERS]) to COVID-19. However little is currently known about SARS-CoV-2 with no established therapy or vaccine.

Lai et al in their 2005 publication showed that "Even with a relatively high virus load (SARS-CoV) in the droplet, rapid loss of infectivity was observed for paper and cotton material" and that "all disinfectants (used in the study) reduced the virus load (SARS-CoV) by 13 log within 5 min after incubation". In addition, it has been shown that viruses (including corona family of viruses) can be de-activated when they come in contact with surfaces covered with sodium chloride (table salt). This can be explained by "physical destruction of virus during recrystallization of coated salts. When the salt-coated fiber is exposed to virus aerosols, salt crystals below the aerosol droplet dissolve to increase osmotic pressure to virus. Due to evaporation, the salt concentration of the droplet significantly increases and reaches the solubility limit, leading to recrystallization of salt. As a consequence, virus particles are exposed to increasing osmotic pressure during the drying process and are physically damaged by crystallization." In 1961, Spier et al showed that viral replication is inhibited by the presence of chloride / halide salts. In addition, a recent report showed that non-myeloid cells (e.g. epithelial, fibroblast and hepatic cells) have an innate immune mechanism, which is augmented in the presence of salt (NaCl). The same report also showed that, in cell culture models, DNA, RNA, enveloped and non-enveloped viruses are all inhibited in the presence of NaCl. The antiviral effect was dependent on the availability of chloride ions (and not sodium ions). In the presence viral infection and the availability of NaCl, cells utilize the chloride ions to produce hypochlorous acid (HOCl). Since HOCl is the active ingredient in bleach, which is known to have an antiviral effect, the mechanism could be augmented by supplying chloride ions through NaCl to treat viral infections. The Edinburgh and Lothians Viral Intervention Study (ELVIS), a pilot RCT of hypertonic saline nasal irrigation and gargling (HSNIG) versus standard care in adults with URTI showed a reduction in the duration of illness by 1.9 days (p = 0.01), less over-the-counter medications use by 36% (p = 0.004), less disease transmission within household contacts by 35% (p = 0.006) and less viral shedding by ≥0.5 log10/day (p = 0.04).

Hypertonic saline (HTS) has also been shown to have anti-inflammatory effects on lung epithelium. In addition, inhaled HTS has been shown to have beneficial effects when used for patients with lung diseases (e.g. cystic fibrosis).

Therefore, the combination of the antiviral properties on surfaces and the anti-inflammatory effects of HTS renders such widely available, affordable and cheap therapy amenable for exploring as potentially beneficial in reducing the severity of lung injury in patients with symptomatic COVID-19 with very minimal risk to the patients.

This proposal aims at testing the effect of spraying the routinely used face masks (or for that matter any material to cover nose and mouth) with HTS on the severity of respiratory symptoms and signs of patients with confirmed COVID-19. In addition, the rate for ICU utilization will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* confirmed diagnosis of COVID-19 by PCR and
* Any of the following

  * cough
  * shortness of breath
  * Respiratory rate more than 20 per minute or
  * oxygen saturation 90% or less on room air

Exclusion Criteria:

* Age younger than 18 years
* Pregnancy
* Participation in other COVID-19 intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of respiratory symptoms | Throughout hospital stay on average 21 days
  Cough and / or shortness of breath
Improvement of respiratory signs | Throughout hospital stay on average 21 days
  Respiratory rate and / or need for supplemental oxygen

SECONDARY OUTCOMES:
ICU admission | Throughout hospital stay on average 21 days
  Rate
Mechanical ventilation | Throughout hospital stay on average 21 days
  Rate

CONTACTS AND LOCATIONS:
Overall Officials: Ali Alshanqeeti, MD, Principal Investigator — King Faisal Specialsit Hospital and Research Center
Locations (1):
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai MY, Cheng PK, Lim WW. Survival of severe acute respiratory syndrome coronavirus. Clin Infect Dis. 2005 Oct 1;41(7):e67-71. doi: 10.1086/433186. Epub 2005 Aug 22. PMID 16142653
- [Background] Quan FS, Rubino I, Lee SH, Koch B, Choi HJ. Universal and reusable virus deactivation system for respiratory protection. Sci Rep. 2017 Jan 4;7:39956. doi: 10.1038/srep39956. PMID 28051158
- [Background] Speir, R. W. (1961). Effect of Several Inorganic Salts on Infectivity of Mengo Virus. Proceedings of the Society for Experimental Biology and Medicine, 106(2), 402-404. https://doi.org/10.3181/00379727-106-26352
- [Background] Ramalingam S, Cai B, Wong J, Twomey M, Chen R, Fu RM, Boote T, McCaughan H, Griffiths SJ, Haas JG. Antiviral innate immune response in non-myeloid cells is augmented by chloride ions via an increase in intracellular hypochlorous acid levels. Sci Rep. 2018 Sep 11;8(1):13630. doi: 10.1038/s41598-018-31936-y. PMID 30206371
- [Background] Ramalingam S, Graham C, Dove J, Morrice L, Sheikh A. A pilot, open labelled, randomised controlled trial of hypertonic saline nasal irrigation and gargling for the common cold. Sci Rep. 2019 Jan 31;9(1):1015. doi: 10.1038/s41598-018-37703-3. PMID 30705369
- [Background] Wright FL, Gamboni F, Moore EE, Nydam TL, Mitra S, Silliman CC, Banerjee A. Hyperosmolarity invokes distinct anti-inflammatory mechanisms in pulmonary epithelial cells: evidence from signaling and transcription layers. PLoS One. 2014 Dec 5;9(12):e114129. doi: 10.1371/journal.pone.0114129. eCollection 2014. PMID 25479425
- [Background] Nydam TL, Moore EE, McIntyre RC Jr, Wright FL, Gamboni-Robertson F, Eckels PC, Banerjee A. Hypertonic saline attenuates TNF-alpha-induced NF-kappaB activation in pulmonary epithelial cells. Shock. 2009 May;31(5):466-72. doi: 10.1097/SHK.0b013e31818ec47d. PMID 18948845
- [Background] Gamboni F, Anderson C, Mitra S, Reisz JA, Nemkov T, Dzieciatkowska M, Jones KL, Hansen KC, D'Alessandro A, Banerjee A. Hypertonic Saline Primes Activation of the p53-p21 Signaling Axis in Human Small Airway Epithelial Cells That Prevents Inflammation Induced by Pro-inflammatory Cytokines. J Proteome Res. 2016 Oct 7;15(10):3813-3826. doi: 10.1021/acs.jproteome.6b00602. Epub 2016 Aug 29. PMID 27529569
- [Background] Mitra S, Schiller D, Anderson C, Gamboni F, D'Alessandro A, Kelher M, Silliman CC, Banerjee A, Jones KL. Hypertonic saline attenuates the cytokine-induced pro-inflammatory signature in primary human lung epithelia. PLoS One. 2017 Dec 18;12(12):e0189536. doi: 10.1371/journal.pone.0189536. eCollection 2017. PMID 29253007
- [Background] Deree J, Martins JO, Leedom A, Lamon B, Putnam J, de Campos T, Hoyt DB, Wolf P, Coimbra R. Hypertonic saline and pentoxifylline reduces hemorrhagic shock resuscitation-induced pulmonary inflammation through attenuation of neutrophil degranulation and proinflammatory mediator synthesis. J Trauma. 2007 Jan;62(1):104-11. doi: 10.1097/TA.0b013e31802d96cb. PMID 17215740
- [Background] Pimentel RN, Petroni RC, Barbeiro HV, Barbeiro DF, Andrade MM, Ariga SK, Soriano FG. Hypertonic solution-induced preconditioning reduces inflammation and mortality rate. J Inflamm (Lond). 2019 Jul 3;16:16. doi: 10.1186/s12950-019-0220-4. eCollection 2019. PMID 31312113
- [Background] Reeves EP, Molloy K, Pohl K, McElvaney NG. Hypertonic saline in treatment of pulmonary disease in cystic fibrosis. ScientificWorldJournal. 2012;2012:465230. doi: 10.1100/2012/465230. Epub 2012 May 3. PMID 22645424
- [Background] Reeves EP, McCarthy C, McElvaney OJ, Vijayan MS, White MM, Dunlea DM, Pohl K, Lacey N, McElvaney NG. Inhaled hypertonic saline for cystic fibrosis: Reviewing the potential evidence for modulation of neutrophil signalling and function. World J Crit Care Med. 2015 Aug 4;4(3):179-91. doi: 10.5492/wjccm.v4.i3.179. eCollection 2015 Aug 4. PMID 26261770
- [Background] Wise SK, Lin SY, Toskala E, Orlandi RR, Akdis CA, Alt JA, Azar A, Baroody FM, Bachert C, Canonica GW, Chacko T, Cingi C, Ciprandi G, Corey J, Cox LS, Creticos PS, Custovic A, Damask C, DeConde A, DelGaudio JM, Ebert CS, Eloy JA, Flanagan CE, Fokkens WJ, Franzese C, Gosepath J, Halderman A, Hamilton RG, Hoffman HJ, Hohlfeld JM, Houser SM, Hwang PH, Incorvaia C, Jarvis D, Khalid AN, Kilpelainen M, Kingdom TT, Krouse H, Larenas-Linnemann D, Laury AM, Lee SE, Levy JM, Luong AU, Marple BF, McCoul ED, McMains KC, Melen E, Mims JW, Moscato G, Mullol J, Nelson HS, Patadia M, Pawankar R, Pfaar O, Platt MP, Reisacher W, Rondon C, Rudmik L, Ryan M, Sastre J, Schlosser RJ, Settipane RA, Sharma HP, Sheikh A, Smith TL, Tantilipikorn P, Tversky JR, Veling MC, Wang Y, Westman M, Wickman M, Zacharek M. International Consensus Statement on Allergy and Rhinology: Allergic Rhinitis. Int Forum Allergy Rhinol. 2018 Feb;8(2):108-352. doi: 10.1002/alr.22073. PMID 29438602
- [Background] Tarrant BJ, Le Maitre C, Romero L, Steward R, Button BM, Thompson BR, Holland AE. Mucoactive agents for chronic, non-cystic fibrosis lung disease: A systematic review and meta-analysis. Respirology. 2017 Aug;22(6):1084-1092. doi: 10.1111/resp.13047. Epub 2017 Apr 11. PMID 28397992
- [Background] Lin L, Chen Z, Cao Y, Sun G. Normal saline solution nasal-pharyngeal irrigation improves chronic cough associated with allergic rhinitis. Am J Rhinol Allergy. 2017 Mar 1;31(2):96-104. doi: 10.2500/ajra.2017.31.4418. PMID 28452705
- [Background] Liedtke CM. Understanding the cellular mechanism for inhaled hyperosmotic saline therapy for patients with cystic fibrosis. Focus on "Effect of apical hyperosmotic sodium challenge and amiloride on sodium transport in human bronchial epithelial cells from cystic fibrosis donors". Am J Physiol Cell Physiol. 2013 Dec 1;305(11):C1096-7. doi: 10.1152/ajpcell.00250.2013. Epub 2013 Aug 28. No abstract available. PMID 23986195
- [Background] Huiberts A, Zweijpfenning SMH, Pennings LJ, Boeree MJ, van Ingen J, Magis-Escurra C, Hoefsloot W. Outcomes of hypertonic saline inhalation as a treatment modality in nontuberculous mycobacterial pulmonary disease. Eur Respir J. 2019 Jul 11;54(1):1802143. doi: 10.1183/13993003.02143-2018. Print 2019 Jul. No abstract available. PMID 31000680